CLINICAL TRIAL: NCT00287898
Title: Telephone-Based Genetic Counseling; An Equivalence Trial
Brief Title: Telephone-Based Genetic Counseling or Standard Genetic Counseling in Women at Risk of Carrying the BRCA1 or BRCA2 Mutation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000450959; R01CA082346 (NIH); R01CA108933 (NIH); P30CA051008 (NIH); GUMC-2004-133
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telephone Genetic Counseling (Experimental): Participants randomized to this arm will receive all genetic counseling via telephone.
  Interventions: Behavioral: Telephone Genetic Counseling
- Usual Care (Active Comparator): Participants randomized to usual care will receive standard in-person genetic counseling.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Telephone Genetic Counseling — Participants will receive all genetic counseling via telephone
  Arms: Telephone Genetic Counseling
Behavioral: Usual Care — subjects will receive standard in-person genetic counseling
  Arms: Usual Care

SUMMARY:
RATIONALE: Genetic counseling may work as well over the telephone as it does in-person. It is not yet known whether genetic counseling by telephone is more effective than standard (in-person) genetic counseling in women at risk of carrying the BRCA1 or BRCA2 mutation.

PURPOSE: This randomized phase III trial is studying telephone-based genetic counseling to see how well it works compared to standard (in-person) genetic counseling in women at risk of carrying the BRCA1 or BRCA2 mutation.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the impact of telephone genetic counseling (TGC) versus standard genetic counseling (SGC) on utilization of BRCA1/BRCA2 testing in women at risk of carrying the BRCA1/BRCA2 mutation.
* Compare the relative efficacy of TGC versus SGC on satisfaction with the counseling process, informed decision making, psychosocial distress, and quality of life.

Secondary

* Identify participant characteristics that predict differential response to TGC.
* Explore the mechanisms by which TGC or SGC impact distress and quality of life.

OUTLINE: This is a randomized, multicenter study. Participants are stratified according to participating site. Participants are randomized to 1 of 2 groups.

* Group 1 (standard genetic counseling): Participants undergo an in-person genetic counseling session. Participants are then given the option of providing blood for genetic testing at the study site. Participants who choose to undergo genetic testing receive their results in-person from their genetic counselor.
* Group 2 (telephone-based genetic counseling): Participants undergo a telephone-based genetic counseling session. Participants who choose to undergo genetic testing receive a pre-labeled blood kit in the mail. Participants receive their results over the phone from their genetic counselor.

After completion of genetic counseling, all participants are followed periodically for 1 year.

PROJECTED ACCRUAL: A total of 600 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Must have at least 10% chance of carrying the BRCA1/BRCA2 gene, as defined by ≥ 1 of the following:

  * First-degree relative of affected family member with a 50% chance of inheriting a BRCA1/BRCA2 mutation
  * Second-degree relative with BRCA1/BRCA2 mutation with 25% risk of inheritance (parent deceased)
  * Obligate gene carrier or affected woman
* Must live within 100 miles of the Lombardi Comprehensive Cancer Center
* No more than 4 weeks since breast or ovarian cancer diagnosis
* No metastatic or inflammatory breast cancer or ovarian cancer
* No stage III breast or ovarian cancer while undergoing concurrent chemotherapy

PATIENT CHARACTERISTICS:

* No psychiatric illness or cognitive disorder that would preclude informed consent

PRIOR CONCURRENT THERAPY:

* No prior genetic counseling or testing for BRCA1 and/or BRCA2

Ages: 21 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 669 (Actual)
Dates: Start 2005-05 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Uptake of BRCA1/BRCA2 mutation testing as measured by genetic test results at 3 and 6 months | 6 months
Knowledge assessed by genetic testing knowledge measure at post-counseling and 3 months | 3 months
Decision making as assessed by Decisional Conflict Satisfaction at post-counseling and 3 months | 3 months
Quality of life as assessed by SF-12 health survey at 3 and 6 months | 6 months
Distress as assessed by Impact of Events Scale Brief Symptom Inventory MICRA at 3 and 6 months | 6 months

SECONDARY OUTCOMES:
Costs by cost measurement post-counseling | 6 months
Management behaviors as assessed by utilization of management options (e.g., mammography, surgery, and chemoprevention) at 6 and 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc Schwartz, PhD, Study Chair — Lombardi Comprehensive Cancer Center
Locations (4):
- United States (4):
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mount Sinai School of Medicine, New York, New York
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont

REFERENCES:
- [Derived] Peshkin BN, Kelly S, Nusbaum RH, Similuk M, DeMarco TA, Hooker GW, Valdimarsdottir HB, Forman AD, Joines JR, Davis C, McCormick SR, McKinnon W, Graves KD, Isaacs C, Garber J, Wood M, Jandorf L, Schwartz MD. Patient Perceptions of Telephone vs. In-Person BRCA1/BRCA2 Genetic Counseling. J Genet Couns. 2016 Jun;25(3):472-82. doi: 10.1007/s10897-015-9897-6. Epub 2015 Oct 12. PMID 26455498
- [Derived] Schwartz MD, Valdimarsdottir HB, Peshkin BN, Mandelblatt J, Nusbaum R, Huang AT, Chang Y, Graves K, Isaacs C, Wood M, McKinnon W, Garber J, McCormick S, Kinney AY, Luta G, Kelleher S, Leventhal KG, Vegella P, Tong A, King L. Randomized noninferiority trial of telephone versus in-person genetic counseling for hereditary breast and ovarian cancer. J Clin Oncol. 2014 Mar 1;32(7):618-26. doi: 10.1200/JCO.2013.51.3226. Epub 2014 Jan 21. PMID 24449235